CLINICAL TRIAL: NCT02711995
Title: Essential Voice Tremor: An Unblinded Crossover Study of Botulinum Toxin Treatment and Injection Augmentation
Brief Title: Essential Voice Tremor: A Study of Botulinum Toxin Treatment and Injection Augmentation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Weill Medical College of Cornell University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 1505016165
Record Dates: First submitted 2016-02-24; First posted 2016-03-17 (Estimated); Results first posted 2018-01-10 (Actual); Last update posted 2018-02-05 (Actual); Status verified 2018-01

CONDITIONS: Essential Tremor
Keywords: botulinum toxin; injection augmentation; essential voice tremor
MeSH Terms: conditions — Essential Tremor | interventions — Botulinum Toxins; Botulinum Toxins, Type A

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- RenuGel (Experimental): Injection augmentation is the injection of a filler material (Brand: RenuGel; generic: Carboxymethylcellulose) into the vocal cords through the skin of the neck, guided by the view from a flexible laryngoscope inserted through the nostril. The flexible laryngoscopy is identical to the procedure that the doctor has used to examine your vocal cords in the past. It is the routine diagnostic evaluation technique of voice disorders.
  Interventions: Drug: RenuGel
- Botulinum toxin (Active Comparator): Botulinum toxin treatment is the injection of botulinum toxin into the muscles of the vocal cords through the skin of the neck. This is identical to the injections you may have received in the past for your disorder.
  Interventions: Drug: Botulinum Toxin

INTERVENTIONS:
Drug: RenuGel — Injection augmentation is the injection of a filler material (Brand: RenuGel; generic: Carboxymethylcellulose) into the vocal cords through the skin of the neck, guided by the view from a flexible laryngoscope inserted through the nostril. The flexible laryngoscopy is identical to the procedure that the doctor has used to examine your vocal cords in the past. It is the routine diagnostic evaluation technique of voice disorders.
  Other Names: generic: Carboxymethylcellulose
  Arms: RenuGel
Drug: Botulinum Toxin — Botulinum toxin treatment is the injection of botulinum toxin into the muscles of the vocal cords through the skin of the neck. This is identical to the injections you may have received in the past for your disorder.
  Other Names: Botox
  Arms: Botulinum toxin

SUMMARY:
Botulinum toxin is the common treatment of choice for patients with Essential Voice Tremor (EVT), but results are not universally beneficial to all patients. Inconsistent results are noted in the literature and are consistent with the PI's clinical experience. Injection augmentation, a well-established treatment for glottic insufficiency, which is a prominent factor in the clinical presentation of Essential Voice Tremor (EVT), has not been studied. By treating patients at separate times with botulinum toxin and injection augmentation in an unblinded prospective crossover treatment study, we can assess functional outcomes of these two treatments with the population of patients with Essential Voice Tremor (EVT).

DETAILED DESCRIPTION:
The purpose of this study is to compare treatment with botulinum toxin to treatment with injection augmentation in patients diagnosed with essential voice tremor.

Botulinum toxin treatment is the injection of botulinum toxin into the muscles of the vocal cords through the skin of the neck. This is identical to the injections you may have received in the past for your disorder.

Injection augmentation is the injection of a filler material into the vocal cords through the skin of the neck, guided by the view from a flexible laryngoscope inserted through the nostril. The flexible laryngoscopy is identical to the procedure that the doctor has used to examine your vocal cords in the past. It is the routine diagnostic evaluation technique of voice disorders.

Periodic injections with botulinum toxin (Botox) is the current standard of care for patients diagnosed with essential voice tremor, but studies show only about 60% of patients benefit substantially enough to continue treatment. Poor vocal fold closure, a common characteristic of essential voice tremor, is treated in other situations (such as vocal fold paralysis or paresis) with injection augmentation; thus there is reason to think that it may be helpful to patients with essential voice tremor, perhaps even to a greater extent than botulinum toxin.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ages 18-100 who have been diagnosed with essential tremor of the voice (EVT) Diagnosis Code 478.75 Laryngeal Spasm.

Exclusion Criteria:

* WCMC subjects under age 18
* Pregnant patients
* Patients with laryngeal pathology besides tremor, including but not limited to polyps and other benign lesions, precancerous or cancerous changes, vocal fold paralysis, or other laryngeal disorders of mobility

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2015-12-15; Primary Completion 2016-09-29 (Actual); Study Completion 2016-09-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lucian Sulica, MD, Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Cornell Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Eight patients were enrolled in the study, and seven patients completed the study. The first participant enrolled on December 15, 2015 and the last patient completed the study on September 29, 2016. All patients were seen at Weill Cornell Medicine ENT located at 1305 York Avenue,5th Floor NY NY 10021
Pre-assignment Details: One patient was excluded prior to the second intervention. Her neurologist started her on a medication that could have confounded our findings, therefore her participation in the study ended. She still received treatment, but was no longer considered a study subject.
Groups:
- Botulinum Toxin First and RenuGel After: Patients with essential voice tremor underwent botulinum toxin chemodenervation injection. After washout (90 days) , patients underwent injection augmentation. Injection augmentation is the injection of a filler material (Brand: RenuGel; generic: Carboxymethylcellulose) into the vocal cords through the skin of the neck, guided by the view from a flexible laryngoscope inserted through the nostril.
Period: First Intervention (30 Days)
Arm/Group | Botulinum Toxin First and RenuGel After
Started | 8
Completed | 8
Not Completed | 0
Period: Washout (90 Days)
Arm/Group | Botulinum Toxin First and RenuGel After
Started | 8
Completed | 7
Not Completed | 1
Not completed — Conflicting medication | 1
Period: Second Intervention (30 Days)
Arm/Group | Botulinum Toxin First and RenuGel After
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Botulinum Toxin First and RenuGel After
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 3
  >=65 years | 4
Age, Continuous [Mean (Full Range); unit: years] | 62 [46 to 82]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7

OUTCOME MEASURES:

1. Primary Outcome: Vocal Tremor Scoring System (VTSS)
Description: The Vocal Tremor Scoring System (VTSS) was developed to standardize the evaluation and scaling of vocal tremor. Tremor at a specific site was scored according to severity by the laryngologist. It can be rated as: none (0), mild/intermittent (1), moderate (2), severe (3). Six different regions were evaluated in this study: base of tongue, larynx, palate, pharyngeal walls, supraglottis, and true vocal folds. The scale range for each region was 0-3. The total score was a summation of all six regions, with a scalar range of 0-18.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
units on a scale
  Base of tongue at Baseline | 0.57 (0.79) | 0.57 (0.53)
  Base of tongue 30 days after intervention | 1 (1.29) | 0.43 (1.13)
  Larynx at Baseline | 1.43 (0.98) | 0.86 (1.46)
  Larynx 30 days after intervention | 1.86 (1.07) | 1.29 (1.25)
  Palate at Baseline | 2.14 (0.9) | 1.71 (0.76)
  Palate 30 days after intervention | 1.71 (0.95) | 1.86 (0.9)
  Pharyngeal walls at baseline | 1.86 (1.35) | 1.86 (0.9)
  Pharyngeal walls 30 days after intervention | 1.86 (0.9) | 1.14 (1.07)
  Supraglottis at Baseline | 2.14 (0.69) | 1.57 (0.98)
  Supraglottis 30 days after intervention | 1 (0.82) | 1.71 (0.76)
  True Vocal Folds at Baseline | 2.14 (0.9) | 1.71 (0.95)
  True Vocal Folds 30 days after intervention | 1.57 (0.98) | 1.43 (1.27)
  Total at Baseline | 10.29 (3.15) | 8.29 (3.25)
  Total at 30 days after intervention | 9 (2.83) | 7.86 (3.98)

2. Secondary Outcome: Acoustic Analysis- Frequencies
Description: For acoustic assessment, subjects produced a sustained /a/ sound at their habitual speaking pitch and loudness and read assessment sentences from the Consensus Audio-Perceptual Evaluation of Voice (CAPE-V)protocol. Tasks were recorded and analyzed using the Analysis of Dysphonia in Speech and Voice (ADSV) and Multi-Dimensional Voice Profile (MDVP) software. A handheld microphone 3 inches from the subjects' mouths was used for all recordings.
  The Sustained Vowel and All-Voiced Sentence protocols of the ADSV were used to obtain cepstral peak prominence fundamental frequency (CPP F0), The MDVP was used to obtain amplitude tremor frequency (Fatr), and fundamental frequency tremor frequency (Fftr).
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: Frequency (Hz)
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
Frequency (Hz)
  CPP F0 Baseline | 203.13 (35.70) | 195.06 (36.15)
  CPP F0 30 Days after Intervention | 194.11 (34.47) | 189.96 (31.27)
  Fatr Baseline | 3.81 (2.21) | 3.69 (1.50)
  Fatr 30 days after intervention | 3.87 (1.05) | 4.09 (0.88)
  Fftr Baseline | 4.53 (1.28) | 4.22 (1.86)
  Fftr 30 days after intervention | 4.11 (1.31) | 4.20 (1.34)

3. Secondary Outcome: Aerodynamic Data- Airflow
Description: Aerodynamic data were collected using the Phonatory Aerodynamic System (PAS) 6600 (Pentax). Subjects held a facemask coupled to a pneumotachometer with a pressure-sensor tube firmly over the nose and mouth, and rested the pressure-sensor tube in the oral cavity above the tongue. They produced sustained /a/ and "We were away a year ago," from which mean airflow wasanalyzed via the Maximum Sustained Phonation and Running Speech protocols.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: Liters per second (L/s)
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
Liters per second (L/s)
  Mean airflow during voicing Baseline | 0.32 (0.47) | 0.34 (0.41)
  Mean airflow during voicing 30 days after interven | 0.38 (0.60) | 0.26 (0.25)
  Mean expiratory airflow Baseline | 0.31 (0.38) | 0.35 (0.40)
  Mean expiratory airflow 30 days after intervention | 0.42 (0.63) | 0.23 (0.21)

4. Secondary Outcome: Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V)
Description: The Consensus Auditory-Perceptual Evaluation of Voice (CAPE-V) is used to describe the severity of auditory-perceptual attributes of a voice problem. It indicates salient perceptual vocal attributes: (a) Overall Severity; (b) Roughness; (c) Breathiness; (d) Strain; (e) Pitch; and (f) Loudness. The CAPE-V displays each attribute accompanied by a 100- millimeter line forming a visual analog scale (VAS). The clinician indicates the degree of perceived deviance from normal for each parameter on this scale, using a tic mark. For each dimension, scalar extremes are unlabeled.
  The scale range is from 0mm to 100mm. Results can indicate distance in mm to describe the degree of deviancy, so the higher the score the more deviancy from the norm there is.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
units on a scale
  Breathiness at Baseline | 40 (31.49) | 47.14 (28.56)
  Breathiness 30 days after intervention | 42.14 (24.3) | 31.43 (27.95)
  Loudness at Baseline | 23.57 (33.26) | 30.71 (31.81)
  Loudness 30 days after intervention | 29.29 (31.01) | 20 (24.32)
  Pitch at Baseline | 45.71 (26.99) | 55.71 (24.57)
  Pitch 30 days after intervention | 41.43 (12.49) | 49.71 (23.75)
  Roughness at Baseline | 32.14 (19.76) | 37.14 (21.38)
  Roughness 30 days after intervention | 32.43 (21.52) | 30.71 (15.39)
  Strain at Baseline | 59.29 (24.4) | 55 (30.41)
  Strain 30 days after intervention | 41.43 (23.22) | 52.86 (23.07)
  Overall at Baseline | 63.71 (24.47) | 64 (27.59)
  Overall after intervention | 55.43 (24.21) | 56.43 (21.93)

5. Secondary Outcome: Voice Handicap Index-10 (VHI-10)
Description: The Voice Handicap Index-10 consists of 10 questions (statements about voice), where patients rate their the frequency of their problems as: never (0), almost never (1), sometimes (2), almost always (3), and always (4). The scores from each answer are added, and can range from 0-40. The higher the score, the worse the patient's perception of their voice handicap.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
units on a scale
  VHI-10 at Baseline | 26.29 (10.69) | 25.86 (10.61)
  VHI-10 at 30 days after Intervention | 23.57 (7.41) | 29.86 (8.49)

6. Secondary Outcome: Percent of Normal Function (PNF)
Description: The Percent of Normal Function (PNF) is a scale for patients to rate their recurrent functions in increments of five, from no function (0%) to normal function (100%). The higher the percentage, the more normal the function as experienced by the patient.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: percentage of normal function
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
percentage of normal function
  PNF at Baseline | 0.40 (0.32) | 0.34 (0.34)
  PNF at 30 days after Intervention | 0.45 (0.23) | 0.44 (0.32)

7. Secondary Outcome: Aerodynamic Data- Peak Air Pressure
Description: Aerodynamic data were collected using the Phonatory Aerodynamic System (PAS) 6600 (Pentax). Subjects held a facemask coupled to a pneumotachometer with a pressure-sensor tube firmly over the nose and mouth, and rested the pressure-sensor tube in the oral cavity above the tongue. A string of five consonant-vowel syllables (/pa/) at a comfortable pitch and loudness were analyzed through the Voicing Efficiency protocol to determine mean peak air pressure.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: Centimeter of water (cm H2O)
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
Centimeter of water (cm H2O)
  Mean peak air pressure Baseline | 6.98 (2.11) | 9.66 (3.97)
  Mean peak air pressure 30 days after intervention | 7.91 (4.13) | 10.08 (4.04)

8. Secondary Outcome: Aerodynamic Data- Loudness
Description: Aerodynamic data were collected using the Phonatory Aerodynamic System (PAS) 6600 (Pentax). Subjects held a facemask coupled to a pneumotachometer with a pressure-sensor tube firmly over the nose and mouth, and rested the pressure-sensor tube in the oral cavity above the tongue. They produced sustained /a/ and "We were away a year ago," from which loudness was analyzed via the Maximum Sustained Phonation and Running Speech protocols.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: Decibel of sound pressure level (dB SPL)
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
Decibel of sound pressure level (dB SPL)
  Mean loudness Baseline | 82.67 (8.26) | 85.16 (5.02)
  Mean loudness 30 Days after Intervention | 81.40 (6.29) | 84.82 (5.04)

9. Secondary Outcome: Aerodynamic Data- Maximum Phonation Time
Description: Aerodynamic data were collected using the Phonatory Aerodynamic System (PAS) 6600 (Pentax). Subjects held a facemask coupled to a pneumotachometer with a pressure-sensor tube firmly over the nose and mouth, and rested the pressure-sensor tube in the oral cavity above the tongue. They produced sustained /a/ from which Maximum Sustained Phonation time was recorded.
Time Frame: Baseline and 30 days after intervention
Measure: Mean (Standard Deviation); unit: seconds (s)
Arm/Group | Botulinum Toxin | RenuGel
Number analyzed (Participants) | 7 | 7
seconds (s)
  Maximum Phonation Time Baseline | 12.27 (10.34) | 10 (10.57)
  Maximum Phonation Time 30 days after intervention | 9.21 (5.08) | 9.34 (7.52)

ADVERSE EVENTS:
Arm/Group | Botulinum Toxin | RenuGel
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes